CLINICAL TRIAL: NCT04293289
Title: Phase 1 Clinical Trial of Boron Neutron Capture Therapy (BNCT) Using CICS-1 and SPM-011 for Malignant Melanoma and Angiosarcoma
Brief Title: Boron Neutron Capture Therapy Using CICS-1 and SPM-011 for Malignant Melanoma and Angiosarcoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Intelligence Care Systems, Inc. (Industry)
Collaborators: Stella Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNCT-001/SPM-011-JAM001
Record Dates: First submitted 2020-02-25; First posted 2020-03-03 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-11

CONDITIONS: Malignant Melanoma; Angiosarcoma
Keywords: BNCT; Boron Neutron Capture Therapy; Borofalan; Melanoma; Angiosacronoma; skin cancer
MeSH Terms: conditions — Melanoma; Hemangiosarcoma; Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Other): BNCT(Boron Neutron Capture Therapy)
  SPM-011 iv administrates at 200 mg/kg/hr for 2 hours before neutron irradiation. During neutoron irradiation with CICS-1, SPM-011 iv continues at 100mg/kg/hr.
  Interventions: Other: CICS-1 (investigational device),SPM-011(investigational drug)

INTERVENTIONS:
Other: CICS-1 (investigational device),SPM-011(investigational drug) — Intravenous administration of SPM-011 and neutron irradiation with CICS-1.

SUMMARY:
Among skin malignancies, patients with malignant melanoma or angiosarcoma are treated with BNCT using CICS-1 and SPM-011 (borofalan (10B)). Through this trial, safety and appropriate treatment dose will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary malignant melanoma or angiosarcoma diagnosed histopathologically
2. Patients with superficial skin lesions whose maximum diameter of the target lesion is 15 cm or less
3. Patients with lesions that are lying 6 cm or less from the skin surface to the deepest part of the tumor
4. Patients with lesions in the head, neck, chest, or extremities
5. Patients who do not have apparent abnormal hematological and biochemical values in the latest screening test within 28 days of registration

Exclusion Criteria:

1. Patients with obvious disseminated lesions
2. Patients who have undergone previous treatment of radiation therapy exceeding 75 Gy for the target lesion.
3. Patients with active lesions / active multiple cancers in addition to the target lesion
4. Patients with infections that require systemic treatment.
5. Patients with active implantable medical devices
6. Patients with a history of BNCT treatment

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The frequency of DLT(Dose Limiting Toxicity) occurence (Safety) | 90 days
  Evaluate the safety at each dose level by the frequency of DLT occurrence

SECONDARY OUTCOMES:
The incidence of adverse events and failures | 180 days
  Evaluate the incidence of adverse events and failures during the study period
Tumor shrinkage ratio, tumor best shrinkage ratio | 30, 60, 90, 180 days
Response rate | 30, 60, 90, 180 days
Progression-free survival | 30, 60, 90, 180 days
Survival length | 30, 60, 90, 180 days
Best response rate for target lesion | 30, 60, 90, 180 days
Progression-free period | 30, 60, 90, 180 days
Period until chronic adverse event | 30, 60, 90, 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center Hospital, Chuo Ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No